CLINICAL TRIAL: NCT05178082
Title: Pre-habilitation Interventions to Empower Patients With Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Geana P Kurita, Senior researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pre-habilitation interventions
Record Dates: First submitted 2021-11-25; First posted 2022-01-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Chronic Non-Cancer Pain
Keywords: Chronic non-cancer pain; Cognitive-behavioral program; Waiting list; Pain catastrophizing; Patient Reported Outcomes

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial for application and assessment of the two interventions. Patients waiting for multidisciplinary pain treatment at Rigshospitalet and Herlev/Gentofte Hospital will be invited to participate and randomly assigned to one of three arms (1:1:1): VP group, ER group or control group (no intervention). Assessments will occur at baseline, 2 months, 6 months, and 12 months after the intervention.
Masking Description: Statistical analysis of data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VP group (Experimental): Participants are linked to online informative videos on chronic pain produced by the Multidisciplinary Pain Centre (Rigshospitalet, DK). Ten video-modules of 2-6 minutes each. 1. Chronic pain development in Denmark, treatment offered at the Centre. 2. How chronic pain can affect life in all its facets. Chronic complex pain explained. 3. Psychological models used to describe affected life domains. The role of dysfunctional thoughts on e.g. anxiety. 4. The connection between pain and factors that can reduce energy level. 5. Pain interference in the familiar dynamic and relations. 6. Information about how to balance activity and rest - and on daily breathing exercises. 7. The Rules and opportunities when health challenges working life e.g. work relocation. 8. The importance of healthy habits regarding eating, sleep, and self-treating. 9. Selection of medication according to the patient's quality of life. 10. Expected side effects of medication and on measures to counteract side effects.
  Interventions: Behavioral: Educational Video-based Pain Program
- ER group (Experimental): Participants will attend a single-session, 2-hour online group class. The program has two main components: didactics and skills acquisition. Participants will learn about pain self-regulation and self-management. The program content includes strategies to empower individuals with chronic non-cancer pain as following: 1) the identification of unhelpful thought patterns in the moment, 2) regulation of cognition and emotion, including thought reframing and mindset, 3) how to decrease physiological hyperarousal using relaxation techniques (binaural relaxation audio file for diaphragmatic breathing and progressive muscle relaxation), and 4) establishing self-soothing actions. At the end of the class, participants will develop a self-tailored plan for implementing these skills/strategies in daily life to use behaviors that modulate attention and counteract helplessness (Darnall et al 2014). The online class will be delivered by a nurse certified in the ER.
  Interventions: Behavioral: Empowered Relief Program
- Control group (No Intervention): Participants in the control group will not receive any of the interventions. This project will not interfere with any current or future pain treatment. After the end of collecting data, the Multidisciplinary Pain Centre will eventually make available the videos that compose VP to all patients.

INTERVENTIONS:
Behavioral: Educational Video-based Pain Program — Educational videos with 10 modules with information about pain.
  Other Names: VP
  Arms: VP group
Behavioral: Empowered Relief Program — Educational online session for skills acquisition to manage pain. Empowered Relief TM by Beth Darnall ©2013-2022 Stanford University
  Other Names: ER
  Arms: ER group

SUMMARY:
The development of alternative methods to address simple clinical needs and easy interventions of self-application are desired in the pre-habilitation period (waiting list). To our knowledge that are very few studies regarding interventions for patients in waiting list for specialized treatment of chronic non-cancer pain (CNCP) and they do not include cognitive-behavioural programs. This project is based on the hypothesis that educational and cognitive-behavioural interventions help to reduce deleterious effects of pain on some areas of patient's life. Therefore, the goal is to test two different interventions to help patients to self-manage their pain and avoid worsening in the pre-clinical period.

DETAILED DESCRIPTION:
It is a randomized controlled trial for application and assessment of two interventions: an educational Video-based Pain Program (VP) and Empowered Relief Program (ER). The primary purpose of our study is to investigate the effect of ER and VP on the Pain Catastrophizing Score in people with CNCP who are waiting for Multidisciplinary pain treatment. The secondary aim is to analyse the effects on other patient reported outcomes such as pain intensity, pain interference in daily activities, pain catastrophizing, pain acceptance, quality of life, mood, perceived change on over-all pain status, as well as consumption of pain medicine and usage of healthcare services. The effects of the two interventions will be compared with each other and a control group.

ELIGIBILITY:
Inclusion Criteria:

* First appointment date at the Multidisciplinary Pain Centre scheduled at least three months after the invitation to participate in this study
* At least 18 years old
* Fluent in the Danish language
* Access to internet
* Willing and available to participate in the study

Exclusion Criteria:

* History of cognitive dysfunction that interfere with understanding of the educational program and answering the questionnaires
* Epilepsy
* Current history of severe depression
* Current use of private pain services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain catastrophizing at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  Pain catastrophizing in the last 24 hours; Pain Catastrophizing Score

SECONDARY OUTCOMES:
Change from baseline pain intensity and interference in daily activities at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  Brief Pain Inventory to measure pain intensity and interference on general activity, mood, walking ability, work, social relations, sleep, and enjoyment of life with other.
Change from baseline pain acceptance at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  Chronic Pain Acceptance Questionnaire to assess engagement in activity (despite pain), pain willingness, and total pain acceptance score.
Change from baseline health status at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  The Measure Yourself Medical Outcome Profile (MYMOP 2), which measures effects on patient self generated outcome on physical, emotional, or social symptoms/problems. It is problem-specific and includes general wellbeing.
Change from baseline health-related quality of life at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  RAND 36-Item Short Form Health Survey version 1.0 to assess physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
Change from baseline anxiety at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  General Anxiety Disorder - 7 (GAD-7) is commonly used as a measure of general anxiety severity.
Change from baseline depression at 2, 6 and 12 months | Baseline, 2 months, 6 months, and 12 months after the intervention
  Patient Health Questionnaires scale (PHQ-9) can help track a patient's overall depression severity as well as track the improvement of specific symptoms with treatment.
Use of medication and health care system at 2, 6 and 12 months | 2 months, 6 months, and 12 months after the intervention
  Medication used (type and quantity), the number of times that he/she used the health care system because of chronic pain problem and treatment received (pharmacologic, surgical, rehabilitation, etc.), and number of absent days at work because of pain.

OTHER OUTCOMES:
Satisfaction with the interventions at 2, 6 and 12 months | 2 months, 6 months, and 12 months after the intervention
  One general question about satisfaction with the intervention used (6-point scale) and additional comments.

CONTACTS AND LOCATIONS:
Overall Officials: Geana Kurita, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, København Ø., Denmark

IPD SHARING:
Plan to Share IPD: No